CLINICAL TRIAL: NCT02669511
Title: Open-label, Non-randomized, Phase 2 Study Evaluating Efficacy and Safety of PQR309 in Patients With Relapsed or Refractory Primary Central Nervous System Lymphoma
Brief Title: PQR309 in Patients With Relapsed or Refractory Primary Central Nervous System Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PIQUR Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQR309-005
Record Dates: First submitted 2016-01-07; First posted 2016-02-01 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: DLBCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- PQR309 (Other): A single arm study with PQR309, a phosphoinositide-3-kinases (PI3K) and inhibitor of the mammalian target of rapamycin (mTOR), 60mg/80mg given once a day, orally.
  Interventions: Drug: PQR309

INTERVENTIONS:
Drug: PQR309 — Oral PQR309, 80mg or 60mg daily or intermittent dosing
  Other Names: bimiralisib

SUMMARY:
An open-label, non-randomized, two-stage, multicenter study evaluating clinical efficacy, safety and pharmacokinetics of PQR309 in patients with relapsed or refractory Primary Central Nervous System Lymphoma (PCNSL).

DETAILED DESCRIPTION:
An open-label, non-randomized, two-stage, multicenter study evaluating clinical efficacy, safety, and pharmacokinetics effects of PQR309 in patients with relapsed or refractory Primary Central Nervous System Lymphoma (PCNSL).

The first stage of the study will enroll a minimum of 12 patients with relapsed or refractory Primary Central Nervous System Lymphoma (PCNSL) evaluable for the primary study objective. If during the first stage of the study data emerge that 80 mg p.o. qd is not adequately tolerated or is inefficacious in patients with relapsed or refractory Primary Central Nervous System Lymphoma (PCNSL), additional patients may be enrolled in the study to evaluate alternative dosing regimens, either a lower daily dose (eg. 60 mg) or a lower weekly dose with administration on 2 consecutive days followed by 5 days without treatment in 7-day treatment cycles (intermittent dosing schedule A).In all cases data from at least 12 evaluable patients will be required on the selected dosing regimen (daily or weekly) before the decision is made to proceed with this regimen into the second stage of the study.Nine (9) additional patients will be enrolled for the second stage of the study, for a minimum of 21 patients on the selected dosing regimen in total, evaluable for the final primary endpoint analysis.All patients evaluable for the primary endpoint will be followed until disease progression or death.

Secondary objectives, PQR309 treatment safety and pharmacokinetics (PK) will be evaluated in all enrolled patients in both study stages.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Patient with histologically/cytologically confirmed Primary Central Nervous System Lymphoma (PCNSL)
3. Relapsed or refractory Primary Central Nervous System Lymphoma (PCNSL) demonstrated by cranial MRI.
4. Presence of at least one lesion of bi-dimensionally measurable disease on baseline
5. MRI with a contrast-enhancing tumor of at least 1 cm (10 mm) in the longest diameter.
6. Maximum one prior systemic therapy regimen.
7. If receiving corticosteroids, patients must have been on a stable or decreasing dose of corticosteroids and no more than 8 mg dexamethasone (or equivalent) for at least 5 days prior to date of enrollment.
8. Karnofsky Performance Score (KPS) ≥ 70%.
9. More than 4 weeks from any investigational agent.
10. Adequate haematological, liver and renal function
11. Able and willing to swallow and retain oral medication.
12. Female and male patients of reproductive potential must agree to use effective contraception from screening until 90 days after discontinuing study treatment.
13. Willing and able to sign the informed consent and to comply with the protocol for the duration of the study.

Exclusion Criteria:

1. Central Nervous System (CNS) Lymphoma or chronic immunosuppression-associated central nervous system (CNS) lymphoma.
2. Previous allogeneic hematopoietic stem cell transplant (HSCT transplant).
3. Previous whole brain radiotherapy (WBRT)
4. Other concomitant anti-tumor therapy as determined by the study team.
5. Patients unable to undergo contrast-enhanced MRI.
6. Prior treatment with a phosphoinositide -3 kinase (PI3K) inhibitor, Protein Kinase B Inhibitor is known as AKT inhibitor, or mammalian target of rapamycin (mTOR) inhibitor.
7. Patient taking enzyme-inducing anti-epileptic drug (EIAED) < 7 days of the first dose of PQR309.
8. Patient is taking a drug with a risk to promote QT prolongation and Torsades de Pointes.
9. Patient is currently using herbal preparations or medications. Patient should stop using herbal medications 7 days prior to the first dose of the study drug.
10. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders.
11. Anxiety ≥ Common Terminology Criteria (CTC) of adverse events (AE) grade 3.
12. Patient has an uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, HIV infection, chronic liver disease.

    chronic renal disease, pancreatitis, chronic pulmonary disease, active cardiac disease or cardiac dysfunction, interstitial lung disease, active autoimmune disease, uncontrolled diabetes, neuropsychiatric or social situations that would limit compliance with the study requirements.
13. Presence of gastrointestinal disease or any other condition that could interfere significantly with the absorption of the study drug.
14. Concomitant treatment with medicinal products that increase the potential hydrogen (pH), reduce acidity of the upper gastrointestinal tract, including, but not limited to, proton-pump inhibitors (e.g. omeprazole), H2-antagonists (e.g. ranitidine) and antacids. Patients may be enrolled in the study after a washout period sufficient to terminate their effect.
15. Patient has a history of invasive malignancy other than Primary Central Nervous System Lymphoma (PCNSL). Patients are eligible, if they are disease-free for at least 3 years and deemed to be at low risk for recurrence by the investigator. Patients diagnosed with cervical cancer in situ, basal cell or squamous cell carcinoma of the skin and treated within the past 3 years are eligible.
16. Women who are pregnant or breast feeding.
17. Women able to conceive and unwilling to practice an effective method of birth control from screening until 90 days after discontinuing study treatment (women of childbearing potential must have a negative serum pregnancy test within 7 days prior to first dose of PQR309).
18. Fasting glucose > 7.0 mmol/L (126 mg/dL). or HbA1c > 6.4%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11-12; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Every 8 weeks up to 6 months
  ORR including complete response (CR, unconfirmed complete(CRu) and partial response (PR) according to the 2005 Response Criteria of the Central Nervous System (CNS) Lymphoma Collaborative Group (IPCG)

SECONDARY OUTCOMES:
Number of adverse events (AE) as related to the study medication. | Week 1 Day 1 to 30 days after last dose up to 12 months
  Continous Dosing and Intermittent Dosing
Changes in puls rate | Week 1 Day 1 prior to treatment, Treatment on Day 8,Day 15 and 22, Day 43 and every subsequent 3 weeks, at the end of treatment and 30days after last dose
  Continous Dosing and Intermittent Dosing
Changes in blood pressure | Week 1 Day 1 prior to treatment, Treatment on Day 8,Day 15 and 22, Day 43 and every subsequent 3 weeks, at the end of treatment and 30days after last dose
  Continous Dosing and Intermittent Dosing
Changes in body weight | Week 1 Day 1 prior to treatment, Treatment on Day 8,Day 15 and 22, Day 43 and every subsequent 3 weeks, at the end of treatment and 30days after last dose
  Continous Dosing and Intermittent Dosing
Changes in temperature | Week 1 Day 1 prior to treatment, Treatment on Day 8,Day 15 and 22, Day 43 and every subsequent 3 weeks, at the end of treatment and 30days after last dose
  Continous Dosing and Intermittent Dosing
Changes in Physical examination according to Karnofsky Performance Status (KPS) | Week 1 Day 1 prior to treatment, Treatment on Day 8,Day 15 and 22, Day 43 and every subsequent 3 weeks, at the end of treatment and 30days after last dose
  Continous Dosing and Intermittent Dosing
Generalized anxiety disorder mood scale score (GAD7) | Treatment on Day 22, Day 43 and every subsequent 3 weeks, at the end of treatment and 30days after last dose
  Continous Dosing and Intermittent Dosing
Depression Test PHQ-9 | Treatment on 22, Day 43 and every subsequent 3 weeks, at the end of treatment and 30days after last dose
  Continous Dosing and Intermittent Dosing
Changes in haematology | Week 1 Day 1 prior to treatment, Treatment on Day 8, Day15,Day 22, Day 36 and Day 43 and every subsequent 3 weeks, at the end of treatment and 30 days after last dose
  Continous Dosing and Intermittent Dosing
Changes in Routine blood chemistry | Week 1 Day 1 prior to treatment, Treatment on Day 8, Day15,Day 22, Day 36 and Day 43 and every subsequent 3 weeks, at the end of treatment and 30 days after last dose
  Continous Dosing and Intermittent Dosing
Changes of Insulin/Glucose/C-Peptide | Week 1 Day 1 prior to treatment, Treatment on Day 8, Day15,Day 22, Day 36 and Day 43 and every subsequent 3 weeks, at the end of treatment and 30 days after last dose
  Continous Dosing and Intermittent Dosing
Changes of haemostasis | Week 1 Day 1 prior to treatment, Treatment on Day 22 and Day 43 and every subsequent 3 weeks, at the end of treatment
  Continous Dosing and Intermittent Dosing
Changes of urinanalysis | Week 1 Day 1 prior to treatment, Treatment on Day 22 and Day 43 and every subsequent 3 weeks, at the end of treatment
  Continous Dosing and Intermittent Dosing
Changes of ECG | Week 1 Day 1 prior to treatment, Treatment on Day 22 and Day 43 and every subsequent 3 weeks, at the end of treatment
  Continous Dosing and Intermittent Dosing

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Korfel, MD, Principal Investigator — Charite-Universitaetsmedizin Berlin (Germany); Uwe Schlegel, Prof, Principal Investigator — Neurologische UniversitätsklinikKnappschaftskrankenhaus Bochum GmbH; Elisabeth Schorb, MD, Principal Investigator — UNIVERSITÄTSKLINIKUM FREIBURGKlinik für Innere Medizin I; Martin Dreyling, Prof, Principal Investigator — Medizinische Klinik und Poliklinik III Klinikum der Universität München; Gerald Illerhaus, Prof, Principal Investigator — Klinik für Hämatologie, Onkologie und PalliativmedizinStuttgart Cancer; Michael Weller, Prof, Principal Investigator — University of Zurich; Daniela Bota, MD, Principal Investigator — Center101 The City Drive SouthOrange, CA 92686

IPD SHARING:
Plan to Share IPD: No